CLINICAL TRIAL: NCT03982355
Title: Development and Validation of a Tumour Oxygenation Monitoring Probe
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 19SM5221
Record Dates: First submitted 2019-05-22; First posted 2019-06-11 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer: Anonymised MRI scans (pre-therapy) of locally advanced breast cancer sufferers.
  Interventions: Device: DRS probe
- Rectal Cancer: Anonymised MRI scans (pre-therapy) of locally advanced rectal cancer sufferers.
  Interventions: Device: DRS probe

INTERVENTIONS:
Device: DRS probe — The Oxygenation measurements of the novel diffuse reflectance spectroscopy probe

SUMMARY:
Laboratory based study in which novel tissue oxygenation probe with the potential provide novel means for assessing response to cancer treatment will be developed and validated.

DETAILED DESCRIPTION:
Tumour hypoxia is feature common to most solid tumours, with significant implications in tumour aggressiveness, metastatic potential and response to therapy. Tumour oxygenation monitoring is likely, therefore, to provide a valuable adjunct in risk stratification and treatment response monitoring.

Diffuse reflectance spectroscopy (DRS) utilises the differing absorption of oxygenated as compared to deoxygenated haemoglobin to provide an accurate measure of tissue oxygenation.

This project aims to develop and validate a tissue oxygenation probe for cancer monitoring. Using the clinical paradigms of rectal and breast cancer, anonymised MRIs of cancer sufferers will guide simulations of tissue optical properties to develop a DRS probe. The 3D reconstructed sans will then be used to 3D print tissue phantom models on which the DRS probe will be validated against reference bench top analysers.

ELIGIBILITY:
Inclusion Criteria:

* MRIs from Breast or Rectal Cancer patients (10 of each)
* Locally advanced Cancers (Stage 2 or 3)
* Patients who went on to receive neoadjuvant chemoradiotherapy.
* Anonymised scans

Exclusion Criteria:

* MRIs from patients under the age of 18, or older than 99 years old will be excluded.
* MRIs from patients who did not receive neoadjuvant therapy for cancer will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pretreatment anonymised MRIs from (locally advanced) breast and rectal cancer sufferers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ara Darzi, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The anonymised scans will be used for this study alone. The participant identifiable data will not be available to our research team, and the scan data will not be made available outside of the research team.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 anonymised MRI scans, including 10 each from the breast and rectal cancer groups. The inclusion and exclusion criteria are provided to a member of the radiology team who selected the appropriate cases, anonymised the MRIs and provided all 20 DICOM files. All cases were therefore appropriate for inclusion from the outset, and therefore there was other significant events.
Units Other Than Participants: MRIs analyses
Groups:
- Breast Cancer (10): Anonymised MRI scans (pre-therapy) of locally advanced breast cancer sufferers.
  DRS probe: The Oxygenation measurements of the novel diffuse reflectance spectroscopy probe
- Rectal Cancer (10): Anonymised MRI scans (pre-therapy) of locally advanced rectal cancer sufferers.
  DRS probe: The Oxygenation measurements of the novel diffuse reflectance spectroscopy probe
Period: Overall Study
Arm/Group | Breast Cancer (10) | Rectal Cancer (10)
Started | 10; 10 MRIs analyses | 10; 10 MRIs analyses
Completed | 10; 10 MRIs analyses | 10; 10 MRIs analyses
Not Completed | 0; 0 MRIs analyses | 0; 0 MRIs analyses

BASELINE CHARACTERISTICS:
Population: 10 each of MRI scans from patients with locally advanced breast and rectal cancer. The MRIs were anonymised, and as such no population information is available
Units Other Than Participants: MRIs
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Cancer | Rectal Cancer | Total
Number analyzed (Participants) | 10 | 10 | 20
Number analyzed (MRIs) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — No information available: please refer to the above Baseline Analysis Population Description | NA (NA) — No information available: please refer to the above Baseline Analysis Population Description | NA (NA) — No information available: please refer to the above Baseline Analysis Population Description
Sex/Gender, Customized [Count of Participants; unit: Participants]
  NA | NA — No information available: please refer to the above Baseline Analysis Population Description | NA — No information available: please refer to the above Baseline Analysis Population Description | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Count of MRIs Successfully Modelled for Oxygen Correlation
Description: Number of MRIs 3D modelled for oxygenation sensor development
  Note: this outcome measure was orginally expressed as "Oxygenation Correlation" though this was modeled and therefore we have expressed it as above
Time Frame: MRIs were 3D modelled - single time point at time of MRI
Population: Scans analysed and segmented to guide the development of the DRS probe
Measure: Count of Units; unit: MRIs analyses
Units Other Than Participants: MRIs analyses
Arm/Group | Breast Cancer (10) | Rectal Cancer (10)
Number analyzed (Participants) | 10 | 10
Number analyzed (MRIs analyses) | 10 | 10
MRIs analyses | 10 | 10

ADVERSE EVENTS:
Time Frame: Not collected. The anonymised MRIs of patients were used. The patients themselves were never included in the study and so not at risk
Description: Only MRIs used, bot patients. Therefore no risk to patients of adverse events
Arm/Group | Breast Cancer (10) | Rectal Cancer (10)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03982355/Prot_SAP_000.pdf